CLINICAL TRIAL: NCT02358200
Title: Phase I Study to Evaluate the Tolerability, Safety and Efficacy of BMN-673 in Combination With Carboplatin and Paclitaxel in Patients With Advanced Solid Tumor Malignancies That Have BRCA Mutations or Triple Negative Metastatic Breast Cancer
Brief Title: Study of BMN-673 With Carboplatin and Paclitaxel in Patients With Advanced BRCA-mutated Solid Tumor or Triple Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding support for the study was terminated
Sponsor: Pamela Munster (Other)
Collaborators: QuantumLeap Healthcare Collaborative (Other)
Responsible Party: Sponsor-Investigator, Pamela Munster, Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14955
Record Dates: First submitted 2015-01-27; First posted 2015-02-06 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Triple Negative Metastatic Breast Cancer; BRCA-mutated Solid Tumor
MeSH Terms: interventions — talazoparib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): BMN-673: Oral, every day, Days 1-21; Carboplatin: intravenous, every week, 750 μg/day; Paclitaxel: intravenous, every week, 0.75 x Maximum Tolerated Dose μg/day
  Interventions: Drug: BMN-673; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: BMN-673
Drug: Carboplatin
Drug: Paclitaxel

SUMMARY:
Open label, non-randomized, dose escalation and expansion Phase Ia/b trial to evaluate the safety of the combination of BMN 673 and carboplatin, and subsequently BMN 673 in combination with paclitaxel and carboplatin to determine the recommended Phase II dose of the combination.

DETAILED DESCRIPTION:
Poly adenosine diphosphate-ribose polymerase (PARP) 1/2 inhibitors are a novel class of anticancer agents that have shown activity in tumors with defects in DNA repair and may induce synthetic lethality in combination with agents that induce DNA damage by preventing DNA repair.

The rationale of this study is to determine whether a DNA damaging agent can potentiate the cell death induced by PARP inhibitors in individuals with tumor that are more susceptible to chemotherapy.

The study will evaluate the potential benefits of BMN 673 in combination with weekly carboplatin in patients with metastatic tumors associated with BRCA germ line mutations or patients with triple negative breast cancer with no known BRCA mutation, subsequently if tolerated, an additional cohort will examine the feasibility of adding paclitaxel to this combination for any solid tumor malignancies with potential benefit to this combination.

This is the first study to evaluate the safety and efficacy of BMN 673 in combination with carboplatin in patients with either BRCA mutations or TNBC. If tolerable paclitaxel will be added to the combination in any solid tumor malignancies with potential benefit to this combination.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years or older with advanced malignancies for which no standard therapy is available.
* Dose Escalation: Patients with any solid tumor malignancies
* Does Expansion:
* Patients with advanced malignancies that have germline and/or somatic BRCA mutations (cohort gBRCA) Or
* Triple negative (TN) metastatic breast cancer without known BRCA mutation (cohort TNBC). Tumors will be considered TN when:
* Estrogen receptor (ER) expression <1%
* Progesterone receptor (PR) expression <1%
* Her2 negative as per the American Society of Clinical Oncology (ASCO) guidelines
* Paclitaxel expansion: any solid tumor malignancy with potential benefit from this combination and paclitaxel (ASP).
* Dose expansion cohort only: Histological or cytological confirmation of advanced unresectable solid tumors for which no standard therapy is available in patients with a known BRCA germline mutation or those with metastatic triple negative breast cancer without known BRCA mutation (see inclusion criteria one for definition of triple negative breast cancer).. For the paclitaxel cohorts, any solid tumors with potential benefit from this combination and paclitaxel.
* Consent to screening tumor biopsy (for accessible tumors when appropriate) [optional in dose escalation, mandatory in dose expansion]
* Part 2 only: Measureable tumor (RECIST1.1)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Adequate organ function:
* Absolute neutrophil count (ANC) ≥ 1.5 X 109/L
* Hemoglobin (Hgb) ≥9.5 g/dL(transfusion before treatment is allowable if more than 3 days prior to study start)
* Platelets (plt) ≥ 100 x 109/L
* Potassium within normal range, or correctable with supplements;
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x Upper Limit Normal (ULN)
* Serum total bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN, or calculated creatinine clearance ≥ 60ml/min
* Females of child-bearing potential (FCBP) must have negative serum pregnancy test within 7 days before starting study treatment and willingness to adhere to acceptable forms of birth control (a physician-approved contraceptive method: oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) for a minimum of 4 weeks following the discontinuation of study treatment.

FCBP is defined as a sexually mature woman who:

* Has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or,
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time during the preceding 12 consecutive months
* Male subjects with female partner of childbearing potential must agree to the use of a physician-approved contraceptive method throughout the course of the study and for a minimum of 4 weeks following the discontinuation of study treatment.
* Ability to take oral medications

Exclusion Criteria:

* Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half-lives or 4 weeks, whichever is shorter, prior to starting study treatment
* Patients must have recovered from side effects from prior cancer-directed therapy to grade 1 or less (unless deemed not clinically significant by study investigator).
* Major surgery ≤ 4 weeks prior to starting study regimen or who have not recovered from surgery.
* Any known unstable angina, significant cardiac arrhythmia, or New York Heart Association (NYHA) class 3 or 4 congestive heart failure.
* History of myocardial infraction (MI) within 6 month prior to starting study treatment.
* Any significant medical condition, laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
* Any condition that confounds the ability to interpret data from the study.
* Symptomatic central nervous system metastases. Subjects with brain metastases that have been previously treated and are stable for 4 weeks are allowed.
* Malabsorption or uncontrolled peptic ulcer disease
* Grade 2 or higher peripheral neuropathy (paclitaxel arm only)
* Known allergic reaction or poor tolerability to PARP inhibitors, carboplatin, or paclitaxel
* Pregnant or breastfeeding
* Known active human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From date of randomization until the date of Initial response to the first documented tumor progression or date of death from any cause, up to 18 months.
  Response rate of combination (BMN 673 + carboplatin) in patients with BRCA germline mutations or triple negative cancer without known BRCA mutations, in solid tumor malignancies with paclitaxel with a 15 patient cohort expansion at the maximum tolerated dose (MTD). Response and progression in this study will be evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.

SECONDARY OUTCOMES:
Intolerable Toxicity | From first dose to 30 day follow up.
  Analyses of adverse events will be performed for all patients having received at least one dose of study drug. The study will use the CTCAE v4.0 for reporting of non-hematologic adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No